CLINICAL TRIAL: NCT06544577
Title: Safety of Elacestrant in the Treatment of Advanced Breast Cancer Patients With ER+/HER2- and ESR1-mutations Who Have Progressed on at Least One Line of Endocrine Therapy: a Prospective, Non-interventional Real-world Study
Brief Title: Safety of Elacestrant in ER+/HER2- and ESR1 Mutations MBC
Status: Recruiting | Type: Observational
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ABC-RWS-01
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: ESR1 Gene Mutation; Advanced Breast Cancer; Safety
MeSH Terms: interventions — elacestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ELacestrant: Subjects in this cohort will receive elacestrant
  Interventions: Drug: ELacestrant

INTERVENTIONS:
Drug: ELacestrant — 345 mg/day once daily oral dosing

SUMMARY:
This study is a prospective non-interventional real-world study enrolling patients with advanced breast cancer who are ER+/HER2- and have ESR1- gene mutations, collecting information on patients' complaints, physical examination, laboratory tests, imaging tests and adverse events to observe the safety of elacestrant treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. must have a histologically or cytologically confirmed diagnosis of breast cancer with evidence of locally advanced disease unsuitable for excision or radical radiotherapy, or evidence of metastatic disease unsuitable for radical treatment.
* 2. female ≥ 18 years of age
* 3. female subjects must be postmenopausal (meeting any of the following criteria is sufficient) a) Has undergone oophorectomy. b) Age ≥ 60 years. c) 40 years old < age ≤ 60 years old with 1 year of menopause. d) Age <60 years and receiving ovarian suppression therapy.
* 4. ER-positive and HER2-negative status and ESR1-mutation positive must be confirmed.
* 5. must have progressed on at least one line of endocrine therapy prior to enrollment, including monotherapy or combination therapy.
* 6. have normal organ function (as assessed by the investigator).

Exclusion Criteria:

* 1. women who are pregnant or breastfeeding
* 2. known difficulties in tolerating oral medications, or conditions that interfere with the absorption of oral medications or allergies to medications and their excitements
* 3. other conditions that make enrollment in the study unsuitable, at the discretion of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced breast cancer with ER+/HER2- and ESR1- gene mutation
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | 6 months
  Percentage of occurrences of adverse events

SECONDARY OUTCOMES:
Serious adverse event rate | 6 months
  Percentage of occurrences of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Qing Qu, Doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Hainan Hospital of Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Boao Research Hospital, Hainan), Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided